CLINICAL TRIAL: NCT04132180
Title: The EXTREMA Trial: The Impact of Early Versus Late Upper Extremity Mobilization After Split Thickness Skin Autograft on Wound Healing in Adult Burn Patients - A Single Center Non-Inferiority Randomized Clinical Trial
Brief Title: Early Versus Late Upper Extremity Mobilization After Autograft
Acronym: EXTREMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Shahriar Shahrokhi, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 009-2018
Record Dates: First submitted 2018-09-20; First posted 2019-10-18 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mobilization (Experimental)
  Interventions: Other: Early Mobilization
- Late mobilization (Active Comparator)
  Interventions: Other: Late Mobilization

INTERVENTIONS:
Other: Early Mobilization — Range of motion exercises of the upper extremity will be performed under the guidance of the physical therapy team starting on post-operative day 1.
  Arms: Early mobilization
Other: Late Mobilization — The patient's grafted upper extremity will be immobilized using an elbow flexion blocking splint until post-operative day 5.
  Arms: Late mobilization

SUMMARY:
Rationale: There is currently no observational study or randomized clinical trial published evaluating the impact of early versus late mobilization in the upper extremity after split thickness skin autograft. As the current post-operative care protocols vary based on physician preference, evidence is needed to optimize post-operative rehabilitation protocols guided by evidence which optimize wound healing, extremity range of motion, graft site pain, as well as minimize risks of complications and length of stay in hospital.

Objective: To determine if early mobilization is non-inferior to late mobilization of the upper extremity after split thickness skin autograft with regards to wound healing measured as percent graft take on post-operative day 5 in adult burn patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older at the time of surgery.
2. Injury: Acute (within 72h of injury) thermal flame or scald burn.
3. Surgery: Skin split-thickness meshed autograft (STSG) applied directly on the wound bed.
4. Location: Upper extremity burn - distal to the axilla and proximal to the wrist.

Exclusion Criteria:

1. Injury: Electrical and chemical burn.
2. Location: Autograft exclusively to the wrist, hand, axilla or non-upper extremity.
3. Patients on vasopressors the day of the operation.
4. Pre-existing comorbidities causing upper extremity mobility restrictions.
5. Patient unable to comply with mobilization protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Wound healing | Post-operative day 5
  Percent graft take

SECONDARY OUTCOMES:
Wound healing | Post-operative day 14
  Percent graft take
Post-operative clinical outcomes | Post-operative day 5 and 14
  Elbow range of motion measured using a goniometer.
Post-operative clinical outcomes | Post-operative day 5 and 14
  Graft site pain measured using visual analogue scale (0 - no pain to 10 - worst possible pain)
Post-operative complications | Acute hospital stay, up to one year
  Local complications (seroma, hematoma, infection, graft loss) and systemic complications (infection, deep vein thrombosis, pulmonary embolism, myocardial infarction, mortality).
Discharge outcome - disposition | Acute hospital stay, up to one year
  Discharge disposition
Discharge outcome - readiness | Acute hospital stay, up to one year
  Timing of readiness for discharge.
Discharge outcome - length of stay | Acute hospital stay, up to one year
  Length of stay in hospital. From date of admission to date of discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada